CLINICAL TRIAL: NCT05256446
Title: AMG 701 Expanded Access Program
Status: No longer available | Type: Expanded Access
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: AMG701 Expanded Access Program
Record Dates: First submitted 2022-02-15; First posted 2022-02-25 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-08

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: AMG 701

SUMMARY:
Expanded access requests for AMG 701 may be considered for adult patients with relapsed and/or refractory multiple myeloma whose disease is in partial response or better after AMG 420 therapy. To request access, use Responsible Party contact information provided in this record.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen